CLINICAL TRIAL: NCT06994871
Title: Effects of Aerobic or Resistance Exercise, or Both on Intrahepatic Lipid in Patients With Metabolic Dysfunction-associated Steatotic Liver Disease: a Randomized Controlled Trial
Brief Title: Effects of Different Exercises on Intrahepatic Lipid in Patients With Metabolic Dysfunction-associated Steatotic Liver Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Yan Bi, Chief Physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-880-03
Record Dates: First submitted 2025-01-05; First posted 2025-05-29 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Metabolic Dysfunction-Associated Steatotic Liver Disease
MeSH Terms: interventions — Exercise; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic exercise (Experimental): The subjects receive aerobic exercise for 12 weeks.
  Interventions: Other: Aerobic exercise
- Resistance exercise (Experimental): The subjects receive resistance exercise for 12 weeks.
  Interventions: Other: Resistance exercise
- combined exercise (Experimental): The subjects receive both aerobic and resistance exercise for 12 weeks.
  Interventions: Other: combined exercise

INTERVENTIONS:
Other: Aerobic exercise — Intensity of exercise：Subjects conduct an aerobic exercise at 40-59% heart rate reserve(HRR).
  Time of aerobic exercise：from 30 to 45 minutes each day, five days a week.
  Arms: Aerobic exercise
Other: Resistance exercise — The resistance exercise was consisted of equipment trainings and body weight trainings. Participants are required to exercise 3 times a week.
  Intensity of equipment trainings: 70% 1-RM. Exercise volume: 15-20 repetitions for a set, from 2 sets to 4 sets gradually.
  Body weight trainings: 15-30 repetitions for a set, from 2 sets to 4 sets gradually.
  Arms: Resistance exercise
Other: combined exercise — Subjects conduct both aerobic and resistance trainings. Details of aerobic training session: Subjects conduct an aerobic exercise at 40-59% heart rate reserve(HRR) from 50-55 minutes each day, 3-4 days a week.
  Details of resistance training session: The resistance exercise was consisted of equipment trainings and body weight trainings. Participants are required to exercise 2 times a week.
  Arms: combined exercise

SUMMARY:
This is a single-center, randomized, parallel controlled study to explore the effects of aerobic exercise, resistance exercise or aerobic combined resistance exercise on liver lipid in patients with MASLD, consisting of a 12-week core study followed by a 12-month extension phase.

DETAILED DESCRIPTION:
This study was a single-center, randomized, parallel controlled clinical study. It conducted a 12-week exercise intervention for patients with MASLD, aiming to explore the effects of different exercise patterns for patients with MASLD. All subjects were randomly assigned to aerobic exercise, resistance exercise or aerobic combined resistance exercise groups. The liver lipid content was evaluated by MRI-PDFF values at baseline and 12 weeks after intervention. Liver function was evaluated by liver transaminase at baseline and 12 weeks after intervention. The degree of liver fibrosis was evaluated by MRE, LSM value and FIB-4 index at baseline and 12 weeks after intervention. The changes of body weight and body fat before and after the intervention were evaluated by Inbody-770, and the changes of muscle mass before and after the intervention were evaluated by DXA. The effects of different exercise methods on metabolic indexes were evaluated by the changes of blood glucose, glycated hemoglobin, insulin and blood lipid before and after the intervention. In addition, after the exercise intervention, this study plans to conduct a 12-month long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Metabolic dysfunction-associated steatotic liver disease pantients with high willingness and compliance;
2. Age: 18-45 years old;
3. BMI: 25-40kg/m2;
4. Liver MRI-PDFF > 10%;
5. Weight change <3% within 3 months before the intervention;
6. Being sedentary (≤60 minutes/week of moderate intensity exercise)
7. Without diabetes, or combined with type 2 diabetes (lifestyle control and glycated hemoglobin ≤7%).

Exclusion Criteria:

1. Patients with a history of excessive alcohol consumption: Excessive alcohol consumption was defined as an average daily consumption of more than 20g of ethanol in women and 30g in men.
2. Other types of chronic liver disease: such as viral hepatitis, cirrhosis, liver cancer, autoimmune liver disease, Wilson's disease, alpha-1 antitrypsin deficiency, hemochromatosis, drug-induced liver disease, etc.
3. Combined with other metabolic diseases: such as type 1 diabetes, hyperthyroidism, hypothyroidism, cushing syndrome, etc.
4. Patients with cardiovascular disease: such as uncontrolled hypertension, acute coronary syndrome, myocardial infarction, severe arrhythmia requiring medical therapy, etc.
5. Patients with cerebrovascular diseases: such as cerebral hemorrhage, ischemic stroke, etc.
6. Patients with the history of biliary obstruction, neuromuscular disease, skeletal deformity, severe osteoporosis, chronic kidney disease, and malignancy.
7. Patients used drugs which may have potential effects on MASLD within 1 year before randomization, including PPAR agonist, SGLT2 inhibitor, GLP1 receptor agonist, insulin, etc.
8. Patients with the history of bariatric surgery, major surgery within 8 weeks before randomization, etc,
9. Patients were enrolled in another clinical trial for the treatment of MASLD or weight loss within 1 year before randomization.
10. Pregnancy, lactation period, or women who plan to pregnant within 6 months before randomization.
11. Patients with mental healthy problems requiring medication.
12. Inability or unwillingness to undergo magnetic resonance imaging, including claustrophobia, implantable cardioverter defibrillators, and pacemakers.
13. Patients cannot complete 12-week exercise plan due to some reasons, such as frequent business trips.
14. After assessment, patients are not suitable or unable to participate in this clinical trial due to personal reasons.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 186 (Estimated)
Dates: Start 2025-03-09 (Actual); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Changes of intrahepatic triglyceride contents | Baseline, 12 weeks
  The changes of intrahepatic triglyceride contents were measured by MRI-PDFF.

SECONDARY OUTCOMES:
Changes of liver transaminase | Baseline, 12 weeks
  The changes of liver transaminase were measured by ALT, AST, γ-GGT, ALP.
Changes of liver fibrosis | Baseline, 12 weeks
  The changes of liver fibrosis were measured by MRE.
Changes of liver fibrosis degree | Baseline, 12 weeks
  The changes of liver fibrosis were measured by LSM.
Changes of FIB-4 index | Baseline, 12 weeks
  The changes of liver fibrosis can be measured by FIB-4 index.
Changes of body weight | Baseline, 12 weeks
  The changes of body weight were measured by InBody-770 equipment.
Changes of body fat | Baseline, 12 weeks
  The changes of body fat were measured by InBody-770 equipment and dual-energy X-ray absorptionmetry.
Changes of muscle mass | Baseline, 12 weeks
  The changes of muscle mass were measured by InBody-770 equipment and dual-energy X-ray absorptionmetry.
Changes of muscle function | Baseline, 12 weeks
  The changes of muscle function were measured by strength test using athletic equipments.
Changes of HbA1c. | Baseline, 12 weeks
  The changes of glucose metabolism indexes were measured by HbA1c.
Changes of blood glucose | Baseline, 12 weeks
  The changes of glucose metabolism indexes were measured by blood glucose.
Changes of blood insulin | Baseline, 12 weeks
  The changes of glucose metabolism indexes were measured by blood insulin.
Changes of lipid metabolism indexes | Baseline, 12 weeks
  The changes of lipid metabolism indexes were measured by triglyceride, total cholesterol, high-density and low-density lipoprotein-cholesterol.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Bi, MD,PhD, Study Director — Nanjing Drum Tower Hospital, Affiliated Hospital of Medical School, Nanjing University
Locations (2):
- China (2):
  - Department of Endocrinology, the Affiliated Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Department of Endocrinology, the Affiliated Drum Tower Hospital of Nanjing University Medical School, Nanjing

IPD SHARING:
Plan to Share IPD: No